CLINICAL TRIAL: NCT04572607
Title: Effect of Avocado Honey (Apis Mellifera) on Anthropometric and Biochemical Parameters in Healthy Subjects: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Marcelo Hernández-Salazar, PhD. Marcelo Hernández-Salazar, Principal investigator, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 19-FaSPyN-SA-25.TP
Record Dates: First submitted 2020-09-09; First posted 2020-10-01 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Healthy Subjects
Keywords: avocado honey; anthropometric parameters; biochemical parameters; natural sweetener

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (13):
- Control group 1 (No Intervention)
- Control group 2 (No Intervention)
- Control group 3 (No Intervention)
- Control group 4 (No Intervention)
- Control group 5 (No Intervention)
- Control group 6 (No Intervention)
- Control group 7 (No Intervention)
- Honey group 1 (Experimental)
  Interventions: Dietary Supplement: The consumption of avocado honey was analyzed
- Honey group 2 (Experimental)
  Interventions: Dietary Supplement: The consumption of avocado honey was analyzed
- Honey group 3 (Experimental)
  Interventions: Dietary Supplement: The consumption of avocado honey was analyzed
- Honey group 4 (Experimental)
  Interventions: Dietary Supplement: The consumption of avocado honey was analyzed
- Honey group 5 (Experimental)
  Interventions: Dietary Supplement: The consumption of avocado honey was analyzed
- Honey group 6 (Experimental)
  Interventions: Dietary Supplement: The consumption of avocado honey was analyzed

INTERVENTIONS:
Dietary Supplement: The consumption of avocado honey was analyzed — The subjects of honey group consumed 25 g of honey each day for 4 weeks.
  Arms: Honey group 1; Honey group 2; Honey group 3; Honey group 4; Honey group 5; Honey group 6

SUMMARY:
Thirteen healthy subjects (5 males; 8 females) ages 25-50 years, with BMI (body mass index): <25 kg/m2 completed the study. The participants were selected randomly, either the control group (n= 7) or honey group (n= 6). Subjects of honey group consumed 25 g of honey each day for 4 weeks.

DETAILED DESCRIPTION:
18 healthy participants (body mass index [BMI] <25 kg/m2) between 25-50 years of age were recruited, of which 13 subjects (male [n=5]) and female [n=8]) completed the study. The participants were allocated randomly either control group (n= 7) or honey group (n= 6). Subjects of honey group consumed 25 g of honey each day for 4 weeks. Participants of both groups did not undergo a special diet regimen, drug therapy, or change in their lifestyle, such as physical exercise, during the period of study. A 3- day food record including two weekdays and one weekend day was used to assess the habitual food intake of the participants prior to initiation of the trial and repeated each week of intervention. Also, dietary intake was calculated using the database Food Processor® (Version. 10.3.0.), including nutritional information of Mexican foods when they weren't on the list.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Female
* Ages 25-50 years,
* BMI (body mass index): under 25 kg per m2.

Exclusion Criteria:

* Not smoker
* Not have an allergy to honey
* Not pregnant,
* Not been previously diagnosed any disease resulting in metabolic disorders
* Not chronically use medications known to affect metabolism
* Not participate in greater than 3 hours of structured exercise per week.
* Female participants that used some kind of contraceptives

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2020-07-18 (Actual)

PRIMARY OUTCOMES:
Subject numbers that experienced a change of glucose level (mg/dL) post-intake of 25 g/day of honey | From the start of treatment (baseline) until 4 weeks
Subject numbers that experienced change of triglycerides levels (mg/dL) post-intake of 25 g/day honey | From the start of treatment (baseline) until 4 weeks
Subject numbers that experienced change of total cholesterol levels (mg/dL) post-intake of 25 g/day honey | From the start of treatment (baseline) until 4 weeks
Subject numbers that experienced change of HDL-cholesterol levels (mg/dL) post-intake of 25 g/day honey | From the start of treatment (baseline) until 4 weeks
Subject numbers that experienced change of LDL-cholesterol levels (mg/dL) post-intake of 25 g/day honey | From the start of treatment (baseline) until 4 weeks
Subject numbers that experienced change of body weight (kg) post-intake of 25 g/day honey. | Frame: from the start of treatment (baseline) until 4 weeks
Subject numbers that experienced change of body fat (%) post-intake of 25 g/day honey | From the start of treatment (baseline) until 4 weeks
Subject numbers that experienced change of waist circumference (cm) post-intake of 25 g/day honey | From the start of treatment (baseline) until 4 weeks
Subject numbers that experienced change of hip circumference (cm) post-intake of 25 g/day honey | From the start of treatment (baseline) until 4 weeks
Subject numbers that experienced change of waist-hip ratio post-intake of 25 g/day honey | From the start of treatment (baseline) until 4 weeks
Subject numbers that experienced change of BMI (weight (kg)/height (m)2) post-intake of 25 g/day honey | From the start of treatment (baseline) until 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo Hernandez Salazar, PhD, Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Facultad de Salud Publica y Nutricion, Monterrey, Nuevo León, Mexico